CLINICAL TRIAL: NCT03749616
Title: Effect of NSAID Use on Pain and Opioid Consumption Following Distal Radius Fracture: A Prospective, Randomized Study
Brief Title: Effect of NSAID Use on Pain and Opioid Consumption Following Distal Radius Fracture
Acronym: Adult NSAID
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Original principal investigator left the institution and investigator replacing him did not have the patient population to enroll as needed.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Daniel London, Assistant Professor, Orthopedic Surgery, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009129
Record Dates: First submitted 2018-09-26; First posted 2018-11-21 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen (Active Comparator): Acetaminophen for pain control with dose and frequency of 325mg 1-2 tablets q4-6h hours as needed, Maximum dose 1000mg. Maximum amount per day: 3g/day.
  Oxycodone 5mg 1-2 tablets q4-6 hours will be available as needed for breakthrough pain.
  Interventions: Drug: Acetaminophen
- NSAID (Experimental): NSAID administered ibuprofen 400-800 mg, up to three times a day and acetaminophen with dose and frequency of 325mg 1-2 tablets q4-6h hours as needed, Maximum dose 1000mg. Maximum amount per day: 3g/day as needed for pain control.
  Oxycodone 5mg 1-2 tablets q4-6 hours will be available for breakthrough pain.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — NSAID Group - will be administered ibuprofen 400-800 mg, up to three times a day as needed for pain control
  Other Names: Motrin; Advil
  Arms: NSAID
Drug: Acetaminophen — Control Group - will be administered acetaminophen for pain control with dose and frequency of 325mg 1-2 tablets q4-6h hours as needed, Maximum dose 1000mg. Maximum amount per day: 3g/day.
  Other Names: tylenol
  Arms: Acetaminophen

SUMMARY:
Non-steroidal anti-inflammatory drugs (NSAIDs), such as ibuprofen, are excellent medications for providing pain control in certain patients. There is some data to suggest that NSAIDs can be used to reduce postoperative pain and narcotic use in patients who had undergone carpal tunnel release. There are mixed results about the effect of bone healing in adult patients with broken bones. The investigators hypothesize that NSAID administration in the acute phase of distal radius fracture healing will be non-inferior for pain control and decrease the use of opioid analgesics compared to patients who take acetaminophen for pain control during this same time period. Furthermore, the investigators hypothesize that patients will have similar or better patient reported outcomes, range of motion, and strength with the administration of NSAIDs.

DETAILED DESCRIPTION:
In the United States, drug overdose deaths and opioid-involved deaths continue to increase, quadrupling since 1999; six out of ten drug overdose deaths involve an opioid. Overdoses from prescription opioids are a driving factor in the 15-year increase in opioid overdose deaths. The amount of prescription opioids sold to pharmacies, hospitals, and doctors' offices has drastically risen, yet there had not been an overall change in the amount of pain that Americans reported. Deaths from prescription opioids-drugs like oxycodone, hydrocodone, and methadone-have more than quadrupled since 1999.

Non-steroidal anti-inflammatory drugs (NSAIDs) have been shown to control both postoperative pain and pain associated with some orthopaedic injuries in children and adults with certain orthopaedic injuries. Further, the use of NSAIDs for pain control has been shown to lessen the use of narcotic pain medications, the adverse effects of which are well known. With the current opioid epidemic, more research is needed to determine strategies to reduce opioid use in patients with orthopaedic injuries. Chapman et al. showed that NSAIDs can be used effectively to reduce postoperative pain and narcotic use in patients who had undergone carpal tunnel release. Although distal radius fractures are one of the most common fractures, no studies have examined the effect of NSAIDs on distal radius fracture pain. The purpose of this study is to compare pain and narcotic pain medication use in patients who have had distal radius fractures in patients who use NSAIDs to those who do not.

To the authors' knowledge, there have been no clinical prospective, randomized studies to evaluate the effect that NSAIDs have on patients with distal radius fractures. The investigators hypothesize that NSAID administration in the acute phase of distal radius fracture healing will be non-inferior for pain control and decrease the use of opioid analgesics compared to patients who take acetaminophen for pain control during this same time period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Distal radius fracture

Exclusion Criteria:

* Contraindication to NSAID use (ie, cannot tolerate, gastritis, ulcers, chronic kidney disease stage 4 or higher, bleeding disorders/thrombocytopenia)
* Inability to take breakthrough medications
* Regular use of NSAIDs
* Regular use of Narcotics
* Open fracture
* Other orthopaedic injuries (polytrauma)
* Pathologic fracture
* Previous injury to the bone
* Pregnant or plan to become pregnant
* Unable to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A London, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Health Care, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Acetaminophen: Acetaminophen will be given to participants for pain control following their injury.
  Acetaminophen: Control Group - will be administered acetaminophen for pain control with dose and frequency of 325mg 1-2 tablets q4-6h hours as needed, Maximum dose 1000mg. Maximum amount per day: 3g/day.
- NSAID: Ibuprofen will be given to participants for pain control following their injury.
  Ibuprofen: NSAID Group - will be administered ibuprofen 400-800 mg, up to three times a day as needed for pain control
Period: Overall Study
Arm/Group | Acetaminophen | NSAID
Started | 14 | 18
Completed | 7 | 10
Not Completed | 7 | 8
Not completed — Lost to Follow-up | 4 | 7
Not completed — Screen Failure | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen | NSAID | Total
Number analyzed (Participants) | 14 | 18 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 9 | 14 | 23
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 3 | 8 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 13 | 17 | 30
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Oxycodone Tablets Used for Breakthrough Pain.
Description: The number and dosing of oxycodone tablets taken per participant for breakthrough pain will be recorded.
Time Frame: 2 weeks
Population: Data were not collected due to 1.) incomplete medication diaries; and 2.) medication diaries not returned by participants.
Measure: Mean (Standard Deviation); unit: oxycodone tablets
Groups:
- Acetaminophen: Acetaminophen will be given to participants for pain control following their injury.
  Acetaminophen: Control Group - will be administered acetaminophen for pain control with dose and frequency of 325mg 1-2 tablets q4-6h hours as needed, Maximum dose 1000mg. Maximum amount per day: 3g/day. Oxycodone 5mg 1-2 tablets q4-6 hours will be available as needed for breakthrough pain.
- NSAID: Ibuprofen will be given to participants for pain control following their injury.
  Ibuprofen: NSAID Group - will be administered ibuprofen 400-800 mg, up to three times a day as needed for pain control. Oxycodone 5mg 1-2 tablets q4-6 hours will be available as needed for breakthrough pain.
Arm/Group | Acetaminophen | NSAID
Number analyzed (Participants) | 7 | 13
oxycodone tablets | 16.71 (12.01) | 9.92 (11.98)

2. Primary Outcome: Intensity of Pain: Visual Analog Scale (VAS)
Description: The patient will be asked to report their pain on a scale of 0 - 10 using the Visual Analog Scale with 0 being no pain and 10 being the worst pain the patient can imagine.
Time Frame: 2 Week, 6 Week, 3 Month, 6 Month and 1 Year Post Surgery
Population: Due to attrition, the number analyzed at each time point is the number of participants who followed up with the research team. A total of 14 participants in the Acetaminophen group, and a total of 18 participants in the NSAID group were analyzed through the various timepoints. Information was captured via a automated Electronic Data Capture program, which resulted in inconsistent follow-up at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acetaminophen | NSAID
Number analyzed (Participants) | 14 | 18
score on a scale
  2 weeks postop: number analyzed (Participants) | 13 | 17
  2 weeks postop | 2.46 (2.07) | 2.05 (2.82)
  6 weeks postop: number analyzed (Participants) | 7 | 8
  6 weeks postop | 1.0 (1.0) | 1.25 (1.75)
  3 months postop: number analyzed (Participants) | 8 | 9
  3 months postop | 0.75 (1.75) | 1.88 (2.08)
  6 months postop: number analyzed (Participants) | 9 | 9
  6 months postop | 0.88 (1.61) | 2.55 (3.12)
  1 year postop: number analyzed (Participants) | 9 | 9
  1 year postop | 1.11 (1.83) | 1.66 (2.91)

3. Primary Outcome: Fractures Fully Healed
Description: Radiographic evidence of boney healing of the distal radius. This outcome measure is reported as the number of participants in each group with fully healed fractures at the designated time point.
Time Frame: 6 weeks post surgery
Population: Due to attrition, the number analyzed at each time point is the number of participants who followed up with the research team
Measure: Count of Participants; unit: Participants
Arm/Group | Acetaminophen | NSAID
Number analyzed (Participants) | 9 | 9
Participants | 9 | 9

4. Secondary Outcome: QuickDASH
Description: The QuickDASH is a subset of 11 items from the 30-item DASH and is a self-reported questionnaire in which the response options are presented as 5-point Likert scales. At least 10 of the 11 items must be completed for a score to be calculated and the scores range from 0 (no disability) to 100 (most severe disability). This score was designed be useful in patients with any musculoskeletal disorder of the upper limb.
Time Frame: 2 Week, 6 Week, 3 Month, 6 Month and 1 Year Post Surgery
Population: Due to attrition, the number analyzed at each time point is the number of participants who followed up with the research team. At the 1-year postoperative mark, although 9 participants in each group followed up, the questionnaires were not completed. Therefore, the number analyzed is listed as '0' for both groups at this time point
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Acetaminophen: Acetaminophen for pain control with dose and frequency of 325mg 1-2 tablets q4-6h hours as needed, Maximum dose 1000mg. Maximum amount per day: 3g/day.
  Oxycodone 5mg 1-2 tablets q4-6 hours will be available as needed for breakthrough pain.
  Acetaminophen: Control Group - will be administered acetaminophen for pain control with dose and frequency of 325mg 1-2 tablets q4-6h hours as needed, Maximum dose 1000mg. Maximum amount per day: 3g/day.
- NSAID: NSAID administered ibuprofen 400-800 mg, up to three times a day and acetaminophen with dose and frequency of 325mg 1-2 tablets q4-6h hours as needed, Maximum dose 1000mg. Maximum amount per day: 3g/day as needed for pain control.
  Oxycodone 5mg 1-2 tablets q4-6 hours will be available for breakthrough pain.
  Ibuprofen: NSAID Group - will be administered ibuprofen 400-800 mg, up to three times a day as needed for pain control
Arm/Group | Acetaminophen | NSAID
Number analyzed (Participants) | 14 | 18
score on a scale
  2 week postop: number analyzed (Participants) | 5 | 8
  2 week postop | 34.54 (11.74) | 43.18 (6.76)
  6 week postop: number analyzed (Participants) | 8 | 9
  6 week postop | 42.61 (9.92) | 47.22 (5.30)
  3 month postop: number analyzed (Participants) | 4 | 6
  3 month postop | 47.16 (2.18) | 48.10 (4.64)
  6 month postop: number analyzed (Participants) | 1 | 2
  6 month postop | 43.18 (0) | 48.86 (4.82)
  1 year postop: number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) - UE (Upper Extremity)
Description: The PROMIS UE is scored using a T-score metric, where the mean of the general population is set to 50 with a standard deviation of 10. The minimum score on the PROMIS UE is 0, indicating the lowest level of upper extremity function, while the maximum score is 100, indicating the highest level of upper extremity function. Higher scores represent better upper extremity function.
Time Frame: 2 Weeks, 6 Weeks, 3 Months, 6 Months and 1 Year post surgery
Population: Due to attrition, the number analyzed at each time point is the number of participants who followed up with the research team. At the 1-year postoperative mark, although 9 participants in each group followed up, the questionnaires were not completed by all participants. Therefore, the number of participants who completed the questionnaires and analyzed is listed as at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acetaminophen | NSAID
Number analyzed (Participants) | 14 | 18
score on a scale
  2 week postop: number analyzed (Participants) | 6 | 8
  2 week postop | 21.37 (3.2) | 31.5 (10.44)
  6 week post: number analyzed (Participants) | 8 | 9
  6 week post | 34.86 (11.12) | 40.81 (11.90)
  3 month postop: number analyzed (Participants) | 4 | 6
  3 month postop | 41.6 (13.57) | 47.35 (9.18)
  6 month postop: number analyzed (Participants) | 1 | 2
  6 month postop | 42.3 (0) | 51.9 (8.91)
  1 year postop: number analyzed (Participants) | 0 | 1
  1 year postop |  | 58.2 (0)

6. Secondary Outcome: Grip Strength
Description: Grip strength refers to the force exerted by your hand muscles when you hold or squeeze something measured in kilograms. It's an essential measure of hand function and overall health. To assess grip strength, you can use a dynamometer-a device that measures the force applied during a handgrip. The test involves squeezing the dynamometer as hard as possible, typically with the elbow bent at a 90-degree angle. Grip strength varies based on factors such as age, sex and hand dominance.
Time Frame: 2 Week, 6 Week and 3 Month Post Surgery
Population: Due to attrition, the number analyzed at each time point is the number of participants who followed up with the research team. Grip Strength testing was not completed by all participants. Therefore, the number of participants who completed grip strength testing and were analyzed is listed as at these time points.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Acetaminophen | NSAID
Number analyzed (Participants) | 13 | 15
kilograms
  2 week postop: number analyzed (Participants) | 0 | 2
  2 week postop |  | 10.67 (9.54)
  6 week postop: number analyzed (Participants) | 8 | 9
  6 week postop | 12.6 (13.26) | 9.86 (8.49)
  3 month postop: number analyzed (Participants) | 5 | 4
  3 month postop | 9.6 (5.73) | 11.0 (8.25)

7. Secondary Outcome: Key Pinch Strength
Description: Key pinch strength, also known as lateral pinch strength, measures the force exerted by the hand and fingers when pinching an object between the thumb and the radial side of the index finger. Normal ranges typically fall between 10 to 20 pounds of force (4.54 to 9.07 kgs).
Time Frame: 2 weeks, 6 weeks, and 3 months post surgery
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Acetaminophen | NSAID
Number analyzed (Participants) | 14 | 18
kilograms
  2 week postop: number analyzed (Participants) | 2 | 5
  2 week postop | 4.5 (3.11) | 3.25 (1.85)
  6 week postop: number analyzed (Participants) | 8 | 9
  6 week postop | 4.74 (3.22) | 5.56 (3.41)
  3 month postop: number analyzed (Participants) | 5 | 4
  3 month postop | 4.44 (2.18) | 4.58 (1.68)

8. Secondary Outcome: Wrist Range of Motion (ROM)
Description: Wrist ROM refers to the ability of the wrist to move in different directions. Normal wrist extension ranges from 70°- 90° resulting in a normal flexion-extension arc of 140-180°. The minimum wrist motion required for daily activities is 60° of extension, 54° of flexion, or approximately a 100° flexion-extension arc.
  ROM can be varied based on factors such as age, sex, and individual anatomy.
Time Frame: 2 weeks, 6 weeks and 3 months post surgery
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Acetaminophen | NSAID
Number analyzed (Participants) | 14 | 18
degrees
  2 weeks postop: number analyzed (Participants) | 2 | 5
  2 weeks postop | 67.5 (38.89) | 67.6 (38.1)
  6 weeks postop: number analyzed (Participants) | 9 | 9
  6 weeks postop | 89.38 (57.53) | 78.89 (43.12)
  3 months postop: number analyzed (Participants) | 7 | 5
  3 months postop | 76.86 (43.83) | 143.75 (29.26)

ADVERSE EVENTS:
Time Frame: 1 year
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information, did not differ from clinicaltrials.gov.
Arm/Group | Acetaminophen | NSAID
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/18
Other Adverse Events (participants affected / at risk) | 0/14 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT03749616/Prot_SAP_000.pdf